CLINICAL TRIAL: NCT02064374
Title: A Phase I, Open Label, Parallel Group, Three Period, Fixed Sequence Crossover Study to Evaluate the Effect of Dolutegravir on Metformin Pharmacokinetics in Healthy Adult Subjects
Brief Title: Effect of Dolutegravir on Metformin Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201167
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Dolutegravir; drug interaction; metformin; pharmacokinetics; healthy volunteers
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Metformin; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): All subjects will be assigned to a single-sequence of three treatment periods without washout. Subjects will receive Metformin immediate release (IR) 500 mg q12h following a moderate fat meal for 5 days (Period 1), followed by Metformin IR 500 mg q12h plus DTG 50 mg q24h following a moderate fat meal for 7 days (Days 1-7 of Period 2), followed by Metformin IR 500 mg q12h following a moderate fat meal (Days 1-10 of period 3).
  Interventions: Drug: Metformin 500 mg q12h; Drug: Dolutegravir 50 mg q24h
- Cohort 2 (Experimental): All subjects will be assigned to a single-sequence of three treatment periods without washout. Subjects will receive Metformin IR 500 mg q12h following a moderate fat meal (Day 1-5 of Period 1), followed by Metformin IR 500 mg q12h plus DTG 50 mg q12h following a moderate fat meal for 7 days (Days 1-7 of Period 2), followed by Metformin IR 500 mg q12h following a moderate fat meal (Days 1-10 of period 3).
  Interventions: Drug: Metformin 500 mg q12h; Drug: Dolutegravir 50 mg q12h

INTERVENTIONS:
Drug: Metformin 500 mg q12h — Metformin will be supplied as 500 mg tablet to be administered orally.
Drug: Dolutegravir 50 mg q24h — Dolutegravir will be supplied as 50 mg tablet to be administered orally. To be taken once a day in the morning in Period 2 (Total daily dose 50 mg per day for Cohort 1 only)
  Arms: Cohort 1
Drug: Dolutegravir 50 mg q12h — Dolutegravir will be supplied as 50 mg tablet to be administered orally. To be taken 50 mg tablets every 12 hours in Period 2 (Total daily dose 100 mg per day for Cohort 2 only).
  Arms: Cohort 2

SUMMARY:
This study will be a phase 1, open label, parallel group, three period crossover study to evaluate the effect of dolutegravir (DTG) on the steady state pharmacokinetics of metformin and on the safety and tolerability of dolutegravir and metformin. Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow up visit 7-14 days after the last dose of study drug. Eligible subjects will be assigned to one of the two treatment cohorts. Subjects will receive metformin 500 milligram (mg) after every 12 hours (q12h) for 5 days in Period 1; metformin 500 mg q12h plus dolutegravir 50 mg after every 24 hours (q24h) (Cohort 1) or 50 mg q12h (Cohort 2) for 7 days in Period 2; and metformin 500 mg q12h for 10 days in Period 3. There will be no washout periods between treatments. All doses of study drug will be taken following a meal. Safety evaluations will be collected during each period. Serial pharmacokinetic (PK) samples will be collected for metformin on the last day of each period and for dolutegravir on the last day of Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and cardiac monitoring]. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (Kg) for males and >=45 Kg for females and body mass index (BMI) within the range 18.5 - 31.0 Kg/m^2 (square meters) (inclusive).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international units per milliliter (MIU/mL) and estradiol <40 picograms (pg)/mL (<147 picomole per liter (pmol/L) is confirmatory]; Child-bearing potential with negative pregnancy test as determined by [serum or urine] human chorionic gonadotropin (hCG) test at screening or prior to dosing AND Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 5 days post-last dose. OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase, alkaline phosphatase and bilirubin <= 1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Pregnant females as determined by positive [serum or urine] hCG test at screening or prior to dosing.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation. Subjects will allergy to tricyclic antidepressants should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Lactating females.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic pressure is outside the range of 45-90 mmHg, or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening electrocardiogram (ECG) (a single repeat is allowed for eligibility determination): Heart rate for males <45 and >110 bpm and females <50 and >100 bpm; PR interval <120 and >220 msec, QRS duration <70 and >120 msec, QTc interval (Bazett) >450 msec. Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization); any clinically significant arrhythmia which, in the opinion of the investigator and GSK Medical Monitor, will interfere with the safety for the individual subject; any conduction abnormality (including but not specific to left or right incomplete bundle branch block, atrioventricular block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, and non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Steady state plasma metformin pharmacokinetics (PK) parameters | Day 5 to Day 22
  PK parameters will include: maximum concentration (Cmax), area under the time-concentration curve over the dosing interval [AUC(0-tau)]
Steady state plasma DTG PK parameters | Day 12 and Day 13
  PK parameters will include: Area under the time-concentration curve over the dosing interval [AUC(0-tau)], apparent clearance following oral dosing (CL/F), concentration at time zero (C0) and maximum concentration (Cmax)
Steady-state plasma metformin PK parameters in Period 2 as compared to those in Period 1 | Day 5 to Day 12
  PK parameters will include: Terminal phase half-life (t1/2) and Apparent clearance following oral dosing (CL/F)

SECONDARY OUTCOMES:
Change from baseline in vital signs | Upto Day 22
  Vital signs will include systolic and diastolic blood pressure and pulse rate.
Number of subjects with adverse events (AEs) | Upto Day 22
  AEs will be assessed throughout the study.
Toxicity grading of clinical laboratory tests | Upto Day 22
  Laboratory assessments will include haematology, clinical chemistry and urinalysis parameters.
Steady-state plasma metformin PK parameters in Period 3 for each cohort | Upto Day 22
  PK parameters will include: Cmax, concentration curve over the dosing interval [AUC(0-tau)], Terminal phase half-life (t1/2) and apparent clearance following oral dosing (CL/F)
Changes in serum creatinine upon dosing and discontinuation of DTG | Upto Day 22
  Serum creatinine change will be calculated from baseline over time in each period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Song IH, Zong J, Borland J, Jerva F, Wynne B, Zamek-Gliszczynski MJ, Humphreys JE, Bowers GD, Choukour M. The Effect of Dolutegravir on the Pharmacokinetics of Metformin in Healthy Subjects. J Acquir Immune Defic Syndr. 2016 Aug 1;72(4):400-7. doi: 10.1097/QAI.0000000000000983. PMID 26974526